CLINICAL TRIAL: NCT00395954
Title: A Study to Determine the Threshold of Lactose Ingestion That Provokes Symptoms in Lactose Intolerant People.
Brief Title: Amount of Lactose Causing Symptoms in Lactose Intolerant People
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Carolyn Burden, University Hospitals of Leicester NHS Trust
Other Study IDs: UHL 10217
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Lactose Intolerance
Keywords: Lactose Intolerance; Lactose; Threshold
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The hypothesis underlying this study is that failure to recognise the role of lactose intolerance among patients has led to inappropriate dietary advice and treatment with drugs that contain lactose as a filler. These failures exacerbate symptoms and lead to the unnecessary use of immune suppressant drugs.

This study will identify the threshold at which symptoms of lactose intolerance develop, to provide appropriate advice and treatment in the management of patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed lactose intolerance demonstrated with a lactose intolerance test.
* Adherence to a lactose free diet for at least four days before the start of the study.

Exclusion Criteria:

* Failure to adhere to a lactose free diet.
* People who are on lactose containing medications.
* Pregnancy.
* Unwillingness to comply with study outline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Mayberry, DSc MD, Principal Investigator — University Hospitals, Leicester